CLINICAL TRIAL: NCT03063671
Title: Effect of Adding Dexmedetomidine, Ketamine and Their Combination to Bupivicaine in Thoracic Epidural Analgesia on Post-mastectomy Pain
Brief Title: Dexmedetomidine,Ketamine and Their Combination to Bupivicaine on Thoracic Epidural Analgesia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shereen Mamdouh, lectruer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 110
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Acute Pain
Keywords: postmastectomy pain
MeSH Terms: conditions — Acute Pain | interventions — Ketamine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- bupivacine group (Active Comparator): preoperative insertion of thoracic epidural at T4-5 and adminstration of 12 ml bupivacine 0.125% as one shot 15 minutes before general anesthesia postoperative analgesia done by infusion of bupivacaine 0.125% (5ml/hour through thoracic epidural catheter for 12 hours).
  Interventions: Drug: Ketamine, bupivacine,dexmedetomidine
- ketamine group (Active Comparator): preoperative insertion of thoracic epidural at T4-5 and adminstration of 12 ml bupivacine 0.125% plus ketamine in a dose 0.5 mg/kg 15 minutes before general anesthesia postoperative analgesia will be preformed by infusion of mixture of (bupivacaine 0.125% plus ketamine 0.5 mg/ml ml) in a rate of 5ml/hour through thoracic epidural catheter for 12 hours
  Interventions: Drug: Ketamine, bupivacine,dexmedetomidine
- dexmedetomidine group (Active Comparator): preoperative insertion of thoracic epidural at T4-5 and adminstration of 12 ml bupivacine 0.125% plus dexmedetomidine in a dose 1 ug/kg 15 minutes before general anesthesia Postoperative analgesia will be performed using infusion of mixture of (bupivacaine 0.125% plus dexmedetomedine 2μg/ ml) in a rate of 5ml/hour through thoracic epidural catheter for 12 hours.
  Interventions: Drug: Ketamine, bupivacine,dexmedetomidine
- ketamine-dexmedetomidine group (Active Comparator): preoperative insertion of thoracic epidural at T4-5 and adminstration of 12 ml bupivacine 0.125% plus both ketamine in a dose 0.3 mg/kg and dexmedetomidine in a dose 0.1 ug/kg 15 minutes before general anesthesia Postoperative analgesia will be performed using infusion of mixture of (bupivacaine 0.125% plus dexmedetomedine 2μg/ ml and and ketamine 0.5 mg/ml) in a rate of 5ml/hour through thoracic epidural catheter for 12 hours.
  Interventions: Drug: Ketamine, bupivacine,dexmedetomidine

INTERVENTIONS:
Drug: Ketamine, bupivacine,dexmedetomidine — thoracic epidural catheter insertion at T4-5

SUMMARY:
This study investigate the effect of addition dexmedetomidine, ketamine or their combination to bupivacaine in thoracic epidural analgesia on acute postoperative pain after breast cancer surgery.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer diagnosed in Egyptian women. Many modalities are used in the treatment of breast cancer including chemotherapy, radiotherapy or surgical intervention. Nowadays, surgical intervention is more conservative.Modified radical mastectomy (MRM) is the standard surgical procedure of choice in these patients. MRM is usually performed under general anesthesia, almost always combining intravenous and inhalational agents.The drawback of general anesthesia includes inadequate pain control due to lack of analgesia, high incidence of nausea and vomiting, stress of anesthesia and surgery, and increasing the length of hospital stay.Post mastectomy pain is a pain which occur following breast cancer procedures, particularly those operations that remove tissues in upper outer quadrant of breast and/or axilla. This pain can be severe enough to cause long term disabilities and interfere with sleep, performance of daily activities. Also, it can seriously affect the patient mood, and social functions.

Thoracic epidural analgesia (TEA) faces growing interest as adjuvant anesthetic and post-operative analgesic regimen. the use of adjuvant drug with local anesthetic is essential as it prolongs the duration of action, gives better success rate and increases patient satisfaction.

Ketamine, an N-methyl-D-aspartate (NMDA) antagonist, not only abolishes peripheral afferent noxious stimulation, but it can also prevent the central sensitization of nociceptors. When added to epidural local anesthetics, ketamine appears to have adjuvant effects. Dexmedetomedine is a selective, α2-adrenoceptor agonist with analgesic potency, sedative properties, and minimal respiratory depression when used as an adjuvant to regional anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for modified radical mastectomy.
* ASA Physical status I, II and III.

Exclusion Criteria:

* Patients' refusal.
* Uncooperative patients & severe psychiatric illness (cannot evaluate their own pain intensity using visual analogue scale (VAS).
* Patients with history of drug allergy.
* severe renal or liver impairment, unstable ischemic heart disease
* Any contraindications to epidural analgesia (coagulopathy, recent -less than 1 week-treatment with thrombolytic or potent antiplatelet drugs as clopidogrel, and local infection).

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
total dose of intravenous morphine consumption in the first 48 hours post operatively | 48 hours postoperative
  total dose of intravenous morphine comsumption

SECONDARY OUTCOMES:
Visual analogue scale | 0, 2,4,6,8,18,36,48 hours
  Visual analogue scale will be assessed at rest and on movement (abduction of the ipsi-lateral arm).
MAP | 0,30,60,120,150 minutes
  mean arterial blood pressure
HR | 0,30,60,120,150 minutes
  heart rate
sedation score | 0, 2,4,6,8,18,36,48 hours
  sedation sore using sedation scale where; 0 = aware - 1 = drowsy - 2 = asleep/easily respond to verbal command - 3 = asleep/difficulty responding to verbal command -4 = asleep/no respond to verbal command

CONTACTS AND LOCATIONS:
Locations (1):
- south Egypt cancer institute, Asyut, Egypt